CLINICAL TRIAL: NCT00003094
Title: Carotenoid-Rich Diet Trial to Reverse CIN II
Brief Title: Carotenoid Rich Diet in Treating Cervical Dysplasia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was halted prematurely, prior to enrollment of first participant
Sponsor: University of California, San Diego (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Prevention
Other Study IDs: UCSD-960928; CDR0000065806 (Registry Identifier: PDQ (Physician Data Query)); NCI-P97-0100
Record Dates: First submitted 1999-11-01; First posted 2004-04-27 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2007-08

CONDITIONS: Cervical Cancer
Keywords: cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

INTERVENTIONS:
Other: preventative dietary intervention

SUMMARY:
RATIONALE: A diet rich in carotenoids may be an effective treatment for cervical dysplasia.

PURPOSE: Randomized phase II trial to study the effectiveness of a carotenoid rich diet in treating patients with cervical dysplasia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether a carotenoid rich diet will cause a significant increase in the regression of disease in patients with grade I or II cervical intraepithelial dysplasia. II. Determine whether the regression of disease in this patient population is reflected in the modulation of intermediate biological markers (viral genome copy number of human papilloma virus (HPV) and HPV E6/E7 expression).

OUTLINE: This is a randomized, controlled study. Patients are randomized to one of two treatment arms. Arm I: Patients receive dietary counseling and eat 5-10 servings of carotenoid rich fruit and vegetables each day for a year. Arm II: Patients receive no counseling and maintain their normal diet. Carotenoid levels, HPV status, progression of cervical dysplasia, and diet (by food frequency checklist and food diary) are monitored in both groups.

PROJECTED ACCRUAL: A total of 240 patients will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven cervical intraepithelial dysplasia, grade CIN II, or CIN I by repeat cytology No invasive carcinoma by Pap smear No positive endocervical curettage

PATIENT CHARACTERISTICS: Age: 18 to 55 (premenopausal) Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No concurrent beta carotene supplements Not pregnant or nursing No prior malignancy

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: At least 6 months since prior cauterization, cryosurgery, laser, or conization of the cervix

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 1997-10

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl L. Rock, PhD, RD, Study Chair — University of California, San Diego
Locations (1):
- University of California San Diego Cancer Center, La Jolla, California, United States

REFERENCES:
- [Background] Rock CL, Michael CW, Reynolds RK, Ruffin MT. Prevention of cervix cancer. Crit Rev Oncol Hematol. 2000 Mar;33(3):169-85. doi: 10.1016/s1040-8428(99)00073-6. PMID 10789491
- [Background] Ferruzzi MG, Sander LC, Rock CL, Schwartz SJ. Carotenoid determination in biological microsamples using liquid chromatography with a coulometric electrochemical array detector. Anal Biochem. 1998 Feb 1;256(1):74-81. doi: 10.1006/abio.1997.2484. PMID 9466800
- [Background] Gamboa-Pinto AJ, Ferruzi MG, Rock CL, et al.: Relationships between plasma and cervical tissue concentrations in young women. FASEB J 12(5 pt 2): A856, 1998.
- [Background] Gamboa-Pinto AJ, Rock CL, Ferruzzi MG, Schowinsky AB, Schwartz SJ. Cervical tissue and plasma concentrations of alpha-carotene and beta-carotene in women are correlated. J Nutr. 1998 Nov;128(11):1933-6. doi: 10.1093/jn/128.11.1933. PMID 9808645
- [Background] Rock CL. Nutritional factors in cancer prevention. Hematol Oncol Clin North Am. 1998 Oct;12(5):975-91. doi: 10.1016/s0889-8588(05)70037-x. PMID 9888017
- [Background] Rock CL. Dietary Reference Intakes, antioxidants, and beta carotene. J Am Diet Assoc. 1998 Dec;98(12):1410-1. doi: 10.1016/S0002-8223(98)00317-4. No abstract available. PMID 9850107
- [Background] Rock CL. Carotenoids: biology and treatment. Pharmacol Ther. 1997 Sep;75(3):185-97. doi: 10.1016/s0163-7258(97)00054-5. PMID 9504139